CLINICAL TRIAL: NCT01179828
Title: Linking Altered Central Pain Processing and Genetic Polymorphism to Drug Efficacy in Chronic Low Back Pain
Brief Title: Linking Altered Central Pain Processing and Genetic Polymorphism to Drug Efficacy in Chronic Low Back Pain (Predictio)
Acronym: Predictio
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: University of Bern (Other); University of Zurich (Other); Aalborg University (Other)
Responsible Party: Dr Med Andreas Siegenthaler, Inselspital Bern
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: KEK 213/09; grant: SPUM no. 33CM30_124117
Record Dates: First submitted 2010-08-10; First posted 2010-08-11 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2016-04

CONDITIONS: Low Back Pain
Keywords: Quantitative sensory testing; Drug efficacy; Low back pain syndrome; Imipramine; Oxycodone; Clobazam; Tolterodine
MeSH Terms: conditions — Low Back Pain | interventions — Oxycodone; Clobazam; Imipramine; Tolterodine Tartrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Active Comparator): Oxycodone 15mg
  Interventions: Drug: Oxycodone 15mg
- 2 (Active Comparator): Clobazam 20mg
  Interventions: Drug: Clobazam
- 3 (Active Comparator): Imipramine 75mg
  Interventions: Drug: Imipramine
- 4 (Placebo Comparator): Tolterodine 1mg
  Interventions: Drug: Tolterodine

INTERVENTIONS:
Drug: Oxycodone 15mg — 15mg single administration p.o.
  Arms: 1
Drug: Clobazam — 20mg single administration p.o.
  Arms: 2
Drug: Imipramine — 75mg single administration p.o.
  Arms: 3
Drug: Tolterodine — 1 mg single administration p.o.
  Arms: 4

SUMMARY:
Drug therapy in patients with chronic low back pain is a major challenge for physicians. One of the problems is the lacking knowledge in prediction of drug efficacy in a chosen patient. Usually one of the classes of pain medication is given to patients with a similar clinical picture, although different pain mechanisms may be responsible for this clinical picture.

Another reason for variable drug efficacy are genetic polymorphisms, this may be the reason why an unique drug produces different responses (from a lacking analgesic effect up to excessive effect or side-effects.

Quantitative sensory testing is a method that documents alterations in the pain perception system. Linking genetic polymorphisms to quantitative sensory testing may give us a tool for anticipation of drug efficacy.

DETAILED DESCRIPTION:
Background

Drug therapy is an essential part of pain treatment. However, only a minor part of pain patients benefits from the available treatments or is able to tolerate the drugs. One important limitation of drug therapy is lack of instruments to predict their effect. Indeed, in clinical practice "classes" of drugs (e.g. antidepressants) are given to "classes" of patients (e.g. neuropathic pain patients). However, within those classes of patients very different pain mechanisms are likely to underlie the pain condition in different patients. If drugs affect part of these mechanisms, they will not work in all patients. Another reason for variability in drug responses is genetic variation leading to a spectrum of different responses to analgesics, from lack of efficacy to exaggerated responses, up to intolerable adverse effects.

Quantitative sensory testing comprises methods that document alterations and reorganization of the nociceptive system. Measuring an abnormal result in a chronic pain patient may provide us with the information that the underlying pain pathways somehow must be altered. An essential question is whether this information can be linked to drug efficacy in a mechanism-based treatment approach. A further important question is whether assessing genetic polymorphisms can explain different drug effects and hence help selecting the appropriate therapeutic strategy for individual patients.

Objective

We will test the hypothesis that there is a correlation between disturbances in specific pain mechanisms as assessed by quantitative sensory tests and analgesic efficacy after single-dose drug administration in patients with chronic low back pain. Genetic factors affecting drug metabolism and pain sensitivity will be analyzed as additional explanatory variables for drug efficacy.

Methods

Quantitative sensory testing: Heat pain threshold and tolerance, Ice water testing with central modulation of nociceptive input (DNIC), electrical pain detection and temporal summation (skin probe), pressure algometry with pain detection and threshold Drugs investigated: Imipramine, Oxycodone, Clobazam Blood samples: pharmacogenetics: Cytochrome variants CYP2D6, CYP2C19, CYP3A4, COMT haplotypes, CGH-1 variants, A118G of mu opioid receptor gene variants pharmacokinetics: kinetics of imipramine and desipramine

ELIGIBILITY:
Inclusion Criteria:

* Low back pain with NRS>2
* Chronic low back pain since more than 6 months

Exclusion Criteria

* pregnancy
* use of pain medication other than paracetamol and ibuprofen in the last 7 days
* suspicion of radicular pain
* suspicion of intervertebral disk herniation
* foraminal intervertebral stenosis
* suspicion of polyneuropathy
* diabetes
* parkinson disease
* alzheimer disease
* glaucoma
* prostata hyperplasia or voiding problems
* known heart rhythm problems
* heart insufficiency NYHA 3-4
* Systemic inflammatory disease
* Ongoing oncologic disease
* drug or alcohol abuse
* Significant depressive disease (BDI-FS>9)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2010-07; Primary Completion 2015-04 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Difference in NRS(pain scale) between measurement after and before drug administration | 07/2012

SECONDARY OUTCOMES:
Patients global impression of change scale after drug administration | 07/2012
Pharmacogenetic variables(see before) | 07/2012
Pharmacokinetics: measure of Imipramine and desipramine blood levels | 07/2012
Reliability of repeated quantitative sensory testing in the same patient | 12/2010

CONTACTS AND LOCATIONS:
Overall Officials: Michele Curatolo, Prof, Study Chair — University Hospital Bern, Switzerland; Andreas Siegenthaler, Dr Med, Study Director — University Hospital Bern, Switzerland; Pascal H Vuilleumier, Dr Med, Principal Investigator — University Hospital Bern, Switzerland
Locations (1):
- Andreas Siegenthaler, Dep. of Anesthesiolgy and Pain Therapy, Bern University Hospital, Switzerland

REFERENCES:
- [Background] Saarto T, Wiffen PJ. Antidepressants for neuropathic pain. Cochrane Database Syst Rev. 2007 Oct 17;2007(4):CD005454. doi: 10.1002/14651858.CD005454.pub2. PMID 17943857
- [Result] Arendt-Nielsen L, Yarnitsky D. Experimental and clinical applications of quantitative sensory testing applied to skin, muscles and viscera. J Pain. 2009 Jun;10(6):556-72. doi: 10.1016/j.jpain.2009.02.002. Epub 2009 Apr 19. PMID 19380256
- [Result] Foulkes T, Wood JN. Pain genes. PLoS Genet. 2008 Jul 25;4(7):e1000086. doi: 10.1371/journal.pgen.1000086. PMID 18654615
- [Result] Curatolo M, Arendt-Nielsen L, Petersen-Felix S. Central hypersensitivity in chronic pain: mechanisms and clinical implications. Phys Med Rehabil Clin N Am. 2006 May;17(2):287-302. doi: 10.1016/j.pmr.2005.12.010. PMID 16616268
- [Result] Markenson JA, Croft J, Zhang PG, Richards P. Treatment of persistent pain associated with osteoarthritis with controlled-release oxycodone tablets in a randomized controlled clinical trial. Clin J Pain. 2005 Nov-Dec;21(6):524-35. doi: 10.1097/01.ajp.0000146215.86038.38. PMID 16215338
- [Derived] Schliessbach J, Siegenthaler A, Butikofer L, Vuilleumier P, Juni P, Arendt-Nielsen L, Curatolo M. Quantitative sensory tests fairly reflect immediate effects of oxycodone in chronic low-back pain. Scand J Pain. 2017 Oct;17:107-115. doi: 10.1016/j.sjpain.2017.07.004. Epub 2017 Aug 9. PMID 28850362
- [Derived] Siegenthaler A, Schliessbach J, Vuilleumier PH, Juni P, Zeilhofer HU, Arendt-Nielsen L, Curatolo M. Linking altered central pain processing and genetic polymorphism to drug efficacy in chronic low back pain. BMC Pharmacol Toxicol. 2015 Sep 16;16:23. doi: 10.1186/s40360-015-0023-z. PMID 26376691